CLINICAL TRIAL: NCT05886790
Title: A Randomized, Open-Label, Parallel-controlled Clinical Study on Booster Immunization of Two COVID-19 Vaccines Constructed From Different Technical Routes Among People Aged 18 Years and Older
Brief Title: A Clinical Trial on Booster Immunization of Two COVID-19 Vaccines Constructed From Different Technical Routes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Collaborators: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other)
Responsible Party: Principal Investigator, Jianying Huang, Principal Investigator, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMMS85-2301
Record Dates: First submitted 2023-05-29; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; vaccine; immunization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In people aged 18 years and older, people were divided into in three groups and vaccinated using three kinds of vaccines:
  1. Test vaccine 1: Prototype and Omicron BA.4/5 Bivalent Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) For Inhalation
  2. Test vaccine 2: Bivalent COVID-19 mRNA Vaccine
  3. Control vaccine: Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) For Inhalation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Ad5-NCO5T-IH (Experimental): Vaccinated using Prototype and Omicron BA.4/5 Bivalent Recombinant COVID-19 Vaccine(Adenovirus Type 5 Vector) For Inhalation
  Interventions: Biological: Prototype and Omicron BA.4/5 Bivalent Recombinant COVID-19 Vaccine(Adenovirus Type 5 Vector) For Inhalation
- 2. mbO5 (Experimental): Vaccinated using Bivalent COVID-19 mRNA Vaccine
  Interventions: Biological: Bivalent COVID-19 mRNA Vaccine
- 3. Ad5-nCoV-IH (Other): Vaccinated using Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) For Inhalation
  Interventions: Biological: Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) For Inhalation

INTERVENTIONS:
Biological: Prototype and Omicron BA.4/5 Bivalent Recombinant COVID-19 Vaccine(Adenovirus Type 5 Vector) For Inhalation — Containing two adenovirus type 5-based vaccines delivering the spike proteins of SARS-CoV-2 wild type and Omicron BA.4/5 mutant, respectively
  Other Names: Ad5-NCO5T-IH
  Arms: 1. Ad5-NCO5T-IH
Biological: Bivalent COVID-19 mRNA Vaccine — Containing two mRNA-based vaccines delivering the spike proteins of SARS-CoV-2 Beta and Omicron BA.4/5 mutant, respectively
  Other Names: mbO5
  Arms: 2. mbO5
Biological: Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) For Inhalation — Containing adenovirus type 5-based vaccine delivering the spike proteins of SARS-CoV-2 wild type
  Other Names: Ad5-nCoV-IH
  Arms: 3. Ad5-nCoV-IH

SUMMARY:
This is an open-label, randomized, parallel-controlled clinical trial conducted in people aged 18 years and older to evaluate the immunogenicity and safety of two SARS-CoV-2 bivalent vaccines constructed by adenovirus type 5-based or mRNA-based technics.

DETAILED DESCRIPTION:
The clinical trial plans to recruit 450 subjects aged 18 years and above with an interval of ≥ 3 months between the previous dose of SARS-CoV-2 vaccine immunization and receive one dose of inhaled prototype strain and omicron BA.4/5 bivalent recombinant SARS-CoV-2 vaccine (adenovirus vector type 5) (Ad5-NCO5T-IH), beta strain and omicron BA.4/5 bivalent SARS-CoV-2 mRNA vaccine (mbO5) or inhaled prototype recombinant SARS-CoV-2 vaccine (adenovirus vector type 5) (Ad5-nCoV-IH) for follow-up until 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 18 and above at the time of screening;
2. Volunteers can provide with informed consent and sign informed consent form (ICF);
3. Have received COVID-19 vaccine, and the interval between the last vaccination ≥ 3 months.

Exclusion Criteria:

1. Those with convulsions, epilepsy, encephalopathy and serious neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating disease, etc.) in the past five years;
2. Those who are allergic to the active ingredient, any inactive ingredient, or substances used in the production process of the research vaccine, or those who are allergic to the similar vaccines previously; Those who have had severe allergic reactions to vaccines in the past (such as acute allergic reactions, angioedema, dyspnea, etc.), and have any previous history of severe allergies to vaccines, foods, drugs, such as: urticaria, anaphylactic shock, skin eczema, allergic dyspnea, angioedema, etc. or a history of asthma;
3. Those who have previously suffered from severe heart diseases such as myocarditis and pericarditis;
4. Those who have experienced vaccination-related hospitalization or emergency care after previous vaccination;
5. Female urine pregnancy test positive or lactating volunteers, volunteers or their partners have not taken effective contraception 2 weeks before screening or have a pregnancy plan within 6 months;
6. Fever, axillary body temperature≥ 37.3°C;
7. Those with suspected symptoms of COVID-19 in the past 3 months (fever, cough, muscle pain, loss of smell or taste, etc.);
8. Investigators judge that they have known or suspected concomitant serious diseases with unstable drug control, including: respiratory diseases, tuberculosis, acute infection or active chronic disease, liver and kidney disease, cardiovascular disease (cardiopulmonary failure), hypertension (systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥100 mmHg), malignant tumors, infectious or allergic skin diseases;
9. No spleen or functional spleen;
10. Thrombocytopenia, bleeding disorders, or other coagulation disorders (which may cause contraindications to intramuscular injection);
11. Immunosuppressant therapy, anti-allergic therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, superficial corticosteroid therapy for acute non-complicated dermatitis) in the past 6 months;
12. Suffering from nasal or oral diseases, such as acute rhinitis (sinusitis), allergic rhinitis, mouth ulcers, throat redness and swelling, etc.;
13. Have received blood products within 3 months prior to receiving the test vaccine;
14. Have received other vaccines or investigational drugs within 1 month prior to receiving the test vaccine;
15. Are receiving anti-tuberculosis treatment;
16. Those with a history of COVID-19 infection in the past 3 months;
17. Those who have a positive test result of the novel coronavirus antigen at the time of screening;
18. Those with positive HIV infection results at screening;
19. Participated in other interventional studies of lipid-containing nanoparticles;
20. According to the judgment of the investigator, due to various medical, psychological, social or other conditions, it is contrary to the trial protocol, or affects the volunteers' signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-29 (Estimated)

PRIMARY OUTCOMES:
Anti-XBB-specific neutralizing antibody | on day 28 post vaccination
  GMT of anti-XBB-specific neutralizing antibody on day 28 post vaccination
The incidence of adverse reactions | within 28 days post vaccination
  The incidence of adverse reactions within 28 days post vaccination

SECONDARY OUTCOMES:
The incidence of adverse reactions | within 30 mins post vaccination
  The incidence of adverse reactions within 30 mins post vaccination
The incidence of adverse event | within 28 days post vaccination
  The incidence of adverse event within 28 days post vaccination
The incidence of SAE and AESI | within 6 months post vaccination
  The incidence of SAE and AESI within 6 months post vaccination
specific neutralizing antibody against XBB and BA.5 variant on 0 and 28 days | on 0, 28 days post vaccination
  The positive conversion rate, GMT and GMI of specific neutralizing antibody against XBB and BA.5 variant on 0 and 28 days
specific neutralizing antibody against XBB and BA.5 variant at 14 days, 3 and 6 months | at 14 days, 3 and 6 months
  The positive conversion rate, GMT and GMI of specific neutralizing antibody against XBB and BA.5 variant from first 90 subjects at 14 days, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Derived] Wu S, Huang J, Wang B, Li J, Wu J, Zhang Z, Luo L, Zhang J, Huo N, Long J, Huang H, Chen Z, Zhang M, Zhao Z, Dan J, Song X, Mao H, Huo S, Yan H, Zhang Y, Wang X, Hou L. Safety and Immunogenicity of aerosolized adenovirus-vectored COVID-19 vaccine and intramuscular mRNA vaccine bivalent boosters: a randomized open-label clinical trial. Nat Commun. 2025 Aug 7;16(1):7281. doi: 10.1038/s41467-025-62698-7. PMID 40775215